CLINICAL TRIAL: NCT01649752
Title: Phase I Study of Role of Stem Cells in Improving Implantation Rates in ICSI Patients
Brief Title: Role of Stem Cells in Improving Implantation Rates in ICSI Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Nawara Mohamed Hashish, Assistant Professor of Obstetrics and Gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stem cells and implantation
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2012-07

CONDITIONS: Assess the Efficacy of Differentiated and Undifferentiated Stem Cell Therapy in Improving Endometrial Receptivity.
Keywords: Stem cells; Uterine cavity; Implantation; ICSI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Differentiated stem cell therapy group (Experimental): After ovum pick-up, MSC differentiated to endometrium is deposited in the uterine cavity.Embryo transfer will be done at day 5 at the blastocyst stage.
  Interventions: Biological: Differentiated stem cells to endometrium is deposited in the uterine cavity through an IUI catheter
- undifferentiated stem cell therapy group (Experimental): Immediately postmenstrual undifferentiated MSC is deposited in the uterine cavity. Ovum pick-up will be done as usual.Embryo transfer will be done at day 5 at the blastocyst stage.
  Interventions: Biological: Undifferentiated MSC is deposited in the uterine cavity through an IUI catheter.
- Control group (No Intervention): ovum pick-up as usual and embryo transfer at day 5 at the blastocyst stage.

INTERVENTIONS:
Biological: Differentiated stem cells to endometrium is deposited in the uterine cavity through an IUI catheter
  Arms: Differentiated stem cell therapy group
Biological: Undifferentiated MSC is deposited in the uterine cavity through an IUI catheter.
  Arms: undifferentiated stem cell therapy group

SUMMARY:
Background:

Improving implantation rates in ICSI cycles has been the focus of research in recent decades. Because success rates is not satisfactory enough especially when transferring good embryos to the uterine cavity and pregnancy does not occur. Trying to improve endometrial receptivity, the investigators have thought about stem cell therapy as stem cells have played a pivotal role in regenerative medicine in many pathologies as myocardial infarction, Diabetes Mellitus and spinal cord injuries.

Garget and Healy reported in 2011 treatment of a case with Asherman's syndrome by administration of bone marrow stem cells in the uterine cavity. Endometrial growth and improved vascularity has been observed by ultrasound follow-up and Doppler study of endometrial blood flow. Endometrial regeneration has been enough to support pregnancy through successful IVF trial.

The investigators have succeeded in previous work to isolate MSC from placental tissue and differentiate it to endometrium-like cells. The investigators compared the differentiation ability of placental derived mesenchymal stem cells (MSC) and Wharton Jelly derived MSC to differentiate to endometrium under 3 different culture conditions: endometrium conditioned medium (ECM), follicular fluid (FF) conditioned medium and medium containing both. The investigators found that placental MSC has better differentiating ability to endometrium especially under culture conditions containing both ECM and FF as evidenced by prominent appearance of glandular pattern and expression of progesterone receptors in differentiated cells.

Therefore the investigators need to direct this study and test the effect of placental derived MSC in improving implantation rates in patients with recurrent implantation failure, unresponsive endometrium to ovulation induction drugs or with endometrial atrophy or advanced maternal age planning for ICSI trial.

Patients and Methods:

60 patients attending Kasr El-Aini assisted reproduction unit and private IVF center will be randomized to three groups by computer generated programs:

The first group, patients randomized to receive differentiated stem cell therapy:

After ovum pick-up, MSC differentiated to endometrium is deposited in the uterine cavity through an IUI catheter. Embryo transfer will be done at day 5 at the blastocyst stage to allow enough time for endometrial regeneration and increased endometrial receptivity.

The second group, patients randomized to receive undifferentiated stem cell therapy:

Immediately postmenstrual undifferentiated MSC is deposited in the uterine cavity through an IUI catheter to allow enough time for the MSC to differentiate as it needs 7-10 days for differentiation. Ovum pick-up will be done as usual while all other steps will be the same including embryo transfer which will be done at day 5.

The third group, control group:

Patients are randomized to receive no stem cell therapy; All ICSI steps from ovulation induction protocol to embryo transfer conditions will be the same for all groups.

Informed consent will be taken from the patients after detailed explanation of all steps of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ICSI candidates with repeated implantation failure and history of development of good embryos in previous ICSI cycles.
* Advanced maternal age above 38 years.
* Poor endometrial response to ovulation induction drugs.
* Endometrial atrophy.

Exclusion Criteria:

* Presence of infection in the form of vaginitis, cervicitis or hydrosalpinx.
* Presence of uterine abnormality as uterine septum.
* Presence of any pathology distorting the uterine cavity as:

submucus polyp or submucus myoma.

* Marked sperm morphology abnormality.
* High FSH > 12 IU.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 6 months
  Comparison of the implantation rates of all groups; the differentiated stem cell group, the undifferentiated stem cell group and the control group to assess the efficacy of differentiated and undifferentiated stem cell therapy in improving endometrial receptivity.

SECONDARY OUTCOMES:
Endometrial volume and vascularity | 6 months
  Doppler study of the endometrial blood flow; the VI, FI and VFI and 3D-US assessment of endometrial volume in all groups at the day of embryo transfer to obtain objective assessment of the effect of differentiated and undifferentiated stem cell therapy on endometrial volume and vascularity in ICSI patients with advanced maternal age or history of repeated implantation failure.

CONTACTS AND LOCATIONS:
Overall Officials: Nawara Mohamed Hashish, MD, Principal Investigator — Assistant Professor of Gynecology and Obstetrics
Locations (1):
- Kasr El-Aini hospital and private IVF center, Cairo, Egypt